CLINICAL TRIAL: NCT00627523
Title: A Two Year Multicentre, Randomized Two Arm Study Of Genotropin Treatment In Very Young Children Born Small For Gestational Age: Early Growth And Neurodevelopment(Egn)
Brief Title: Genotropin Treatment In Very Young Children Born Small For Gestational Age
Acronym: EGN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A6281287; 2007-003949-32 (EudraCT Number); SGA (Other: Alias Study Number)
Record Dates: First submitted 2008-02-22; First posted 2008-03-03 (Estimated); Results first posted 2014-09-18 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Infant, Small for Gestational Age
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): The active treatment arm
  Interventions: Drug: Genotropin (PN-180,307) Somatropin
- Control (Experimental): Control
  Interventions: Drug: Control-no treatment

INTERVENTIONS:
Drug: Genotropin (PN-180,307) Somatropin — Injectable Genotropin
  Arms: Active
Drug: Control-no treatment — Control-no treatment
  Arms: Control

SUMMARY:
To demonstrate the effect on height and psychomotor development of Growth Hormone treatment in very young children starting at an age of 2 years.

ELIGIBILITY:
Inclusion Criteria:

Caucasian male or female subjects aged between 19-29 months at Screening Visit 1.

Born SGA (birth length and/or weight <-2 SD for gestational age, using country-specific standards).

Height below -2.5 SD at screening (19-29 months of age). At least one measurement of length between 12 and 18 months of age. Normal karyotype in girls to exclude Turners syndrome.

Exclusion Criteria:

Severe Intra-Uterine Growth Retardation (IUGR) (birth length below - 4 SD for gestational age), if associated with dysmorphic features.

Severe prematurity (Gestational Age (GA) <32 weeks of gestation). Ongoing catch-up growth (defined as growth velocity SDS at inclusion >0) based on at least 4 months measurement interval).

Severe familial short stature defined as: Father's height below 155 cm or mother's height below 145 cm.

Defined neurological defects and/or severe neurodevelopmental delay.

Ages: 19 Months to 29 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2008-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- Belgium (2):
  - Universitair Ziekenhuis Brussel/Pediatrie, Brussels
  - Universitair Ziekenhuis Antwerpen / Pediatrie, Edegem
- Czechia (3):
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Ostrava, Detska klinika, Ostrava-Poruba
  - Fakultni nemocnice v Motole, Prague
- CHU Toulouse, Hôpital des Enfants, Service Endocrinologie, Toulouse, France
- Universitaetsklinikum Erlangen, Kinder- und Jugendklinik, Erlangen, Germany
- Italy (4):
  - Centro di Endocrinologia Pediatrica, Dipartimento di Pediatria, Catania
  - Policlinico Universitario, Istituto di Clinica Pediatrica, Messina
  - Dipartimento Materno Infantile, UO di Pediatria e Neonatologia, Milan
  - Dipartimento di Medicina Pediatrica, UO di Endocrinologia e Diabetologia, Roma
- Sophia Children's Hospital, Rotterdam, Netherlands
- Spain (3):
  - Consorci Hospitalari Parc Tauli, Sabadell, Barcelona
  - Hospital Virgen Del Camino, Pamplona, Navarre
  - Hospital Miguel Servet, Zaragoza, Zaragoza
- Drottning Silvias Barn och Ungdomssjukhus, Gothenburg, Sweden
- Inselspital, Ch-3010 Bern, Switzerland

REFERENCES:
- [Derived] De Schepper J, Vanderfaeillie J, Mullis PE, Rooman R, Robertson A, Dilleen M, Gomez R, Wollmann HA. A 2-year multicentre, open-label, randomized, controlled study of growth hormone (Genotropin(R)) treatment in very young children born small for gestational age: Early Growth and Neurodevelopment (EGN) Study. Clin Endocrinol (Oxf). 2016 Mar;84(3):353-60. doi: 10.1111/cen.12968. Epub 2015 Nov 25. PMID 26501737
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6281287&StudyName=Genotropin%20Treatment%20In%20Very%20Young%20Children%20Born%20Small%20For%20Gestational%20Age

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This randomized controlled trial enrolled small for gestational age (SGA) children at 16 centers in 8 countries. In total, 52 participants were screened for the study, of these, 9 participants were considered screen failures. The remaining 43 participants were randomized to receive either study drug (Genotropin®) or were not treated (Control).
Pre-assignment Details: Participants aged between 19 to 29 months at Screening visit, born SGA (birth length and/or weight <-2 standard deviations (SD) for gestational age, using country-specific standards), height below -2.5 SD at Screening (19-29 months of age), and had at least one measurement of length between 12 and 18 months of age were enrolled in this study.
Groups:
- Genotropin®: Participants received Genotropin® at a dose of 0.035 mg/kg/d for 24 months. The dose was calculated based on the actual body weight, and the closest dosing step of the 5 mg pen used. The starting dose for the first 2 weeks was 1/3 of the calculated dose. After 2 weeks the dose was increased to 2/3 of the calculated dose. After 4 weeks the daily dose was the dose calculated on body weight at randomization.
- Control: This group was the untreated control group and was not administered placebo.
Period: Overall Study
Arm/Group | Genotropin® | Control
Started | 21 (22 assigned to Genotropin and 21 in Control; 1 did not take Genotropin, so considered as Control.) | 22
Completed | 19 | 20
Not Completed | 2 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Genotropin® | Control | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Standard Deviation); unit: Months] | 24.91 (3.262) | 24.44 (3.324) | 24.67 (3.263)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Height Standard Deviation Score (SDS) at Month 24.
Description: Height SDS was calculated at the relevant visit by means of the following formula: Height SDS = (participant height) - (normal height)/normal height standard deviation. Where participant height refers to the participant's height at the relevant visit, and normal height and the normal height standard deviation equals the population mean and standard deviation values for participants of a similar age and gender. The change from Baseline value for height SDS was calculated as the difference between the parameter values at a specific visit, and the Baseline parameter values. The scores were centred around zero. Negative score indicated a participant was smaller for their age/gender.
Time Frame: Baseline and Month 24
Population: Full Analysis Set (FAS) included participants who were randomized to treatment and completed at least one post-baseline efficacy measure. Missing values were imputed using LOCF method. One participant was randomized to Genotropin® but did not receive any treatment. This participant was excluded from FAS but included in Control for safety analysis.
Measure: Least Squares Mean (Standard Error); unit: SDS
Arm/Group | Genotropin® | Control
Number analyzed (Participants) | 21 | 21
SDS | 1.63 (0.13) | 0.43 (0.13)
Statistical Analysis 1: Comparison: Genotropin® vs Control; The null hypothesis was that there was no difference in the mean change from Baseline after 24 months in height SDS between the Genotropin® and the untreated control groups. The alternative hypothesis was that there was a difference between the treatment groups; Test type: Superiority or Other; p < 0.001, ANCOVA — ANCOVA model, fitting treatment as a factor, and the baseline parameter value as covariate was used. All hypotheses were tested at a 5% level of significance; No adjustments were made for multiple comparisons; Mean Difference (Final Values) = 1.20, 95% CI 2-sided [0.82 to 1.59], Standard Error of Mean 0.19

2. Secondary Outcome: Change From Baseline in Growth Velocity SDS at Month 24.
Description: The growth velocity SDS was calculated at the relevant visit by means of the following formula: Growth velocity SDS = (participant growth velocity) - (normal growth velocity)/normal growth velocity standard deviation. Where, participant growth velocity refers to the participant's growth velocity at the relevant visit, and normal growth velocity and the normal growth velocity standard deviation equals the population mean and standard deviation values for participants of a similar age and gender. The change from Baseline value for growth velocity SDS was calculated as the difference between the parameter values at a specific visit, and the Baseline parameter values. A negative score indicated that a participant had slower growth for their age/gender.
Time Frame: Baseline and Month 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: SDS
Arm/Group | Genotropin® | Control
Number analyzed (Participants) | 21 | 21
SDS | 0.74 (0.57) | -0.03 (0.57)
Statistical Analysis 1: Comparison: Genotropin® vs Control; The null hypothesis was that there was no difference between the Genotropin® and the untreated control group in terms of the relevant secondary endpoints. The alternative hypothesis was that a difference existed; Test type: Superiority or Other; p = 0.348, ANCOVA — [p-value comment as in outcome 1, analysis 1]; No adjustments were made for multiple comparisons; Mean Difference (Final Values) = 0.77, 95% CI 2-sided [-0.87 to 2.42], Standard Error of Mean 0.81

3. Secondary Outcome: Change From Baseline in Height SDS at Month 12.
Description: as for outcome 1
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: SDS
Arm/Group | Genotropin® | Control
Number analyzed (Participants) | 21 | 21
SDS | 1.03 (0.12) | 0.14 (0.12)
Statistical Analysis 1: Comparison: Genotropin® vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; No adjustments were made for multiple comparisons; Mean Difference (Final Values) = 0.89, 95% CI 2-sided [0.55 to 1.23], Standard Error of Mean 0.17

4. Secondary Outcome: Change From Baseline in Growth Velocity SDS at Month 12.
Description: as for outcome 2
Time Frame: Baseline and Month 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: SDS
Arm/Group | Genotropin® | Control
Number analyzed (Participants) | 21 | 21
SDS | 1.65 (0.56) | -1.59 (0.56)
Statistical Analysis 1: Comparison: Genotropin® vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; No adjustments were made for multiple comparisons; Mean Difference (Final Values) = 3.24, 95% CI 2-sided [1.63 to 4.85], Standard Error of Mean 0.80

5. Secondary Outcome: Change From Baseline in Mental Development Using the Mental Development Index (MDI) of Bayley Scale at Month 12.
Description: The Bayley Scale of Infant Development (BSID-II) measured the mental and psychomotor development and test behavior of participants from 1 to 42 months of age. The scale was used to describe the current developmental functioning of infants and to assist in diagnosis and treatment planning for infants with developmental delays or disabilities. The BSID-II provided the mental raw score which was used to calculate the MDI score. Possible MDI scores ranged from 50-150. A score of 69 and below indicates significantly delayed performance, 70 to 84 indicates mildly delayed performance, 85 to 114 indicates normal limits and 115 and above indicates accelerated performance.
Time Frame: Baseline and Month 12
Population: Full Analysis Set (FAS) included participants who were randomized to treatment and completed at least one post-baseline efficacy measure. One participant was randomized to Genotropin® but did not receive any treatment. This participant was excluded from FAS but included in Control group for safety analysis.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Genotropin® | Control
Number analyzed (Participants) | 21 | 21
Units on a scale | 10.97 (5.34) | 8.55 (4.74)
Statistical Analysis 1: Comparison: Genotropin® vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.738, ANCOVA — ANCOVA model, fitting treatment as a factor, and the baseline parameter value, age, and gender as covariates were used. All hypotheses were tested at a 5% level of significance; No adjustments were made for multiple comparisons; Mean Difference (Final Values) = 2.43, 95% CI 2-sided [-12.27 to 17.12], Standard Error of Mean 7.19

6. Secondary Outcome: Change From Baseline in Psychomotor Development Using the Psychomotor Development Index (PDI) of Bayley Scale at Month 12.
Description: BSID-II measured the mental and psychomotor development and test behavior of participants from 1 to 42 months of age. The scale was used to describe the current developmental functioning of infants and to assist in diagnosis and treatment planning for infants with developmental delays or disabilities. The BSID-II provided the psychomotor raw score which was used to calculate the PDI score. Possible PDI scores ranged from 50-150. A score of 69 and below indicates significantly delayed performance, 70 to 84 indicates mildly delayed performance, 85 to 114 indicates normal limits and 115 and above indicates accelerated performance.
Time Frame: Baseline and Month 12
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Genotropin® | Control
Number analyzed (Participants) | 21 | 21
Units on a scale | 4.04 (3.04) | 8.55 (2.84)
Statistical Analysis 1: Comparison: Genotropin® vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.301, ANCOVA — [p-value comment as in outcome 5, analysis 1]; No adjustments were made for multiple comparisons; Mean Difference (Final Values) = -4.51, 95% CI 2-sided [-13.27 to 4.26], Standard Error of Mean 4.27

7. Secondary Outcome: Head Circumference SDS at Months 3, 6, 12, 18 and 24.
Description: Head circumference SDS was calculated by means of the following formula = (Participant head circumference)-(Normal head circumference)/ Normal head circumference standard deviation. Where participant head circumference refers to the participant's head circumference at the relevant visit, and normal head circumference and the normal head circumference standard deviation equals the population mean and standard deviation values for participants of a similar age and gender. A negative score indicated a participant had a smaller head circumference for their age/gender.
Time Frame: Months 3, 6, 12, 18 and 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Genotropin® | Control
Number analyzed (Participants) | 21 | 21
SDS
  Month 3 (n = 21, 19) | -0.93 (1.217) | -1.37 (1.122)
  Month 6 (n = 21, 19) | -1.20 (1.310) | -1.72 (1.077)
  Month 12 (n = 20, 18) | -0.87 (1.330) | -1.84 (1.158)
  Month 18 (n = 20, 19) | -0.56 (1.890) | -1.76 (1.153)
  Month 24 (n = 20, 20) | -0.75 (1.384) | -1.65 (1.227)

8. Secondary Outcome: Change From Baseline in Head Circumference SDS at Months 3, 6, 12, 18 and 24.
Description: Head circumference SDS was calculated by means of the following formula = (Participant head circumference)-(Normal head circumference)/Normal head circumference standard deviation. Where participant head circumference refers to the participant's head circumference at the relevant visit, and normal head circumference and the normal head circumference standard deviation equals the population mean and standard deviation values for participants of a similar age and gender. A negative score indicated a participant had a smaller head circumference for their age/gender.
Time Frame: Baseline, Months 3, 6, 12, 18 and 24.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Genotropin® | Control
Number analyzed (Participants) | 21 | 21
SDS
  Month 3 (n = 21, 19) | 0.27 (0.977) | 0.36 (0.693)
  Month 6 (n = 21, 19) | -0.00 (0.423) | 0.07 (0.495)
  Month 12 (n = 20, 18) | 0.26 (0.516) | 0.02 (0.587)
  Month 18 (n = 20, 19) | 0.57 (1.094) | 0.04 (0.506)
  Month 24 (n = 20, 20) | 0.39 (0.638) | 0.08 (0.602)

9. Secondary Outcome: Change From Baseline in Body Weight at Months 3, 6, 12, 18, and 24.
Description: Body weight was measured at all the relevant visits. The change from Baseline in body weight was calculated as the difference between the parameter values at each visit, and the Baseline parameter values.
Time Frame: Baseline, Months 3, 6, 12, 18, and 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Genotropin® | Control
Number analyzed (Participants) | 21 | 21
Kg
  Month 3 (n = 21, 19) | 0.57 (0.154) | 0.53 (0.406)
  Month 6 (n = 21, 20) | 1.08 (0.269) | 1.01 (0.659)
  Month 12 (n = 20, 19) | 2.34 (0.389) | 1.66 (0.397)
  Month 18 (n = 20, 19) | 3.48 (0.669) | 2.41 (0.709)
  Month 24 (n = 20, 20) | 4.79 (0.814) | 3.19 (0.601)

10. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at Months 3, 6, 12, 18, and 24.
Description: Body mass index was calculated for all visits by means of the following formula: BMI (kg/m2) = Weight (kg)/(Height[m])2. The change from Baseline BMI was calculated as the difference between the parameter values at each visit, and the Baseline parameter values.
Time Frame: Baseline, Months 3, 6, 12, 18, and 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Kg/m2
Arm/Group | Genotropin® | Control
Number analyzed (Participants) | 21 | 21
Kg/m2
  Month 3 (n = 21, 19) | -0.28 (0.419) | -0.05 (0.811)
  Month 6 (n = 21, 20) | -0.57 (0.537) | 0.08 (1.013)
  Month 12 (n = 20, 19) | -0.62 (0.650) | -0.29 (0.683)
  Month 18 (n = 20, 19) | -0.78 (0.930) | -0.25 (0.806)
  Month 24 (n = 20, 20) | -0.58 (0.823) | -0.55 (0.776)

ADVERSE EVENTS:
Time Frame: Up to the participant's age of 49 to 55 months (Follow-up visit)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Genotropin® | Control
Serious Adverse Events (participants affected / at risk) | 6/21 | 2/22
Other Adverse Events (participants affected / at risk) | 21/21 | 18/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Genotropin® (N=21) | Control (N=22)
Conductive deafness (Ear and labyrinth disorders) | 2 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Hordeolum (Infections and infestations) | 1 | 0
Rotavirus infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Genotropin® (N=21) | Control (N=22)
Ear disorder (Ear and labyrinth disorders) | 1 | 0
Tympanic membrane disorder (Ear and labyrinth disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Regurgitation (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 4
Injection site bruising (General disorders) | 1 | 0
Irritability (General disorders) | 1 | 0
Pyrexia (General disorders) | 9 | 4
Hypersensitivity (Immune system disorders) | 1 | 0
Milk allergy (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 6 | 6
Bronchopneumonia (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 3 | 1
Exanthema subitum (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 2 | 2
Gastroenteritis viral (Infections and infestations) | 2 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 1
Hordeolum (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 4 | 0
Molluscum contagiosum (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 8 | 6
Otitis media (Infections and infestations) | 3 | 1
Otitis media acute (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 2 | 1
Pharyngotonsillitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 2 | 2
Scarlet fever (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 8 | 1
Varicella (Infections and infestations) | 4 | 1
Viral infection (Infections and infestations) | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Growing pains (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchial dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 1
Lipoatrophy (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Haematoma (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.